CLINICAL TRIAL: NCT07352137
Title: Endoscopic Nipple-Sparing Mastectomy (E-NSM) With Immediate Multistage Autologous Fat Grafting(IMAFG) for Total Breast Reconstruction Via the Axillary Incision
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Xue Song, Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZF202418003
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Breast Reconstruction
Keywords: Endoscopic; Nipple-Sparing Mastectomy; Fat Grafting; Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic nipple-sparing mastectomy (E-NSM) with immediate multistage fat grafting (IMFG) (Experimental): Patients with clinical stage 0 to II breast cancer underwent endoscopic nipple-sparing mastectomy (E-NSM) , lymph node surgery, and immediate multistage fat grafting (IMFG) reconstruction using a small cosmetic axillary incision for breast cancer treatment in a single Institution.
  Interventions: Procedure: endoscopic nipple-sparing mastectomy (E-NSM) with immediate implant-based reconstruction

INTERVENTIONS:
Procedure: endoscopic nipple-sparing mastectomy (E-NSM) with immediate implant-based reconstruction — The patient was positioned supine, with the operative-side arm wrapped and elevated to expose the axillary fossa endoscopically. After SLN excision and frozen-section analysis, the lateral edge of the pectoralis major was exposed. A sterile glove finger was used to sheath a wound retractor.Using the electrosurgical hook, the retromammary fat was dissected from the pectoralis major to a defined boundary, carefully preserving the serratus anterior fascia laterally and inferolaterally. Dissection then continued along the marked lateral margin. Subcutaneous breast dissection proceeded with Peng's dissector until the nipple base was transected and sent for frozen section.Fat was harvested via tumescent liposuction from the abdomen or thighs, manually centrifuged, and loaded into 10-mL syringes. It was then injected through the axillary incision into the intramuscular, intermuscular, and submuscular planes of the serratus anterior and pectoralis major muscles.

SUMMARY:
The goal of this clinical study is to evaluate the effectiveness and safety of a novel breast reconstruction technique combining endoscopic nipple-sparing mastectomy (E-NSM) with immediate multistage fat grafting (IMFG) in female patients aged 18 years or older with clinical stage 0 to II breast cancer who desire immediate breast reconstruction. The main questions it aims to answer are:

Does the combined E-NSM and IMFG approach improve patient-reported outcomes, including satisfaction with breasts and physical well-being, as measured by the BREAST-Q questionnaire?

What is the frequency and nature of surgical complications associated with this technique, such as wound healing, hemorrhage, and need for reoperation?

Participants will undergo endoscopic nipple-sparing mastectomy with lymph node surgery followed by immediate multistage fat grafting for total breast reconstruction via a small cosmetic axillary incision. They will also complete the BREAST-Q questionnaire and receive clinical and photography-based assessments at follow-up visits to evaluate aesthetic and quality-of-life outcomes.

ELIGIBILITY:
Inclusion Criteria: • Age >18 years, female

* Stage 0-II( pTis,cT1-2N0-1M0）
* Candidate for a endoscopic nipple- sparing mastectomy procedure (multiple or extensive lesions)
* Patients' choice to undergo an immediate breast reconstruction
* Lack of serious comorbidities
* Accept standard adjuvant therapy

Exclusion Criteria:

* Breast cancer in pregnancy, tumours abutting the chest wall, skin (including inflammatory breast cancer), or nipple-areolar complex (NAC) (including Paget's disease), patients with breast cancer diagnosed as T3 or N2 and above, Allergic to lidocaine

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2027-01-13 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Quality of life(QoL) | 12 months
  QoL at 12 months after the final surgery. The BREAST-Q , version 2.0,22 which was used for measuring pre- and post reconstrucution, has several domains, 3 of which are evaluated for QOL.
The BREAST-Q score | 12months
  Quality of life at 12 months after the final surgery. The BREAST-Q , version 2.0,22 which was used for measuring pre- and post reconstrucution, has several domains, 3 of which are evaluated for QOL: psychosocial well-being, sexual well-being, physical well-being: chest

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial Hospital Of Chinese Medicine, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Result] Lai HW, Chen DR, Liu LC, Chen ST, Kuo YL, Lin SL, Wu YC, Huang TC, Hung CS, Lin YJ, Tseng HS, Mok CW, Cheng FT. Robotic Versus Conventional or Endoscopic-assisted Nipple-sparing Mastectomy and Immediate Prosthesis Breast Reconstruction in the Management of Breast Cancer: A Prospectively Designed Multicenter Trial Comparing Clinical Outcomes, Medical Cost, and Patient-reported Outcomes (RCENSM-P). Ann Surg. 2024 Jan 1;279(1):138-146. doi: 10.1097/SLA.0000000000005924. Epub 2023 May 25. PMID 37226826
- [Result] Zhou J, Xie Y, Liang F, Feng Y, Yang H, Qiu M, Zhang Q, Chung K, Dai H, Liu Y, Liang P, Du Z. A novel technique of reverse-sequence endoscopic nipple-sparing mastectomy with direct-to-implant breast reconstruction: medium-term oncological safety outcomes and feasibility of 24-h discharge for breast cancer patients. Int J Surg. 2024 Apr 1;110(4):2243-2252. doi: 10.1097/JS9.0000000000001134. PMID 38348883
- [Result] Narui K, Satake T, Ishikawa T, Muto M, Tsunoda Y, Yamada A, Kawashima K, Uenaka N, Fujiwara Y, Oshi M, Adachi S, Suzuki C, Wada T, Yamamoto S, Tanabe M, Maegawa J, Endo I. Endoscopic mastectomy followed by immediate breast reconstruction with fat grafting for breast cancer. Breast Cancer. 2024 May;31(3):476-484. doi: 10.1007/s12282-024-01561-x. Epub 2024 Mar 21. PMID 38512534
- [Result] Piatkowski AA, Wederfoort JLM, Hommes JE, Schop SSJ, Krastev TK, van Kuijk SMJ, van der Hulst RRWJ; Breast Reconstruction With External Preexpansion & Autologous Fat Transfer vs Standard Therapy (BREAST) Trial Investigators. Effect of Total Breast Reconstruction With Autologous Fat Transfer Using an Expansion Device vs Implants on Quality of Life Among Patients With Breast Cancer: A Randomized Clinical Trial. JAMA Surg. 2023 May 1;158(5):456-464. doi: 10.1001/jamasurg.2022.7625. PMID 36857058